CLINICAL TRIAL: NCT06462781
Title: Intra-Arterial Injection of Lidocaine and Glucocorticoid in the Treatment of Intractable Headaches: A Non-Randomized, Open-Label Phase 1 Clinical Trial
Brief Title: Localized Injection of Lidocaine and Glucocorticoid for Headache Treatment Phase 1
Acronym: LIGHT 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Collaborators: Society of Vascular and Interventional Neurology (Unknown)
Responsible Party: Principal Investigator, Daniel A Tonetti, MD, Director, Cerebrovascular Neurosurgery; Director, Acute Stroke and NeuroInterventional Suite, The Cooper Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-267
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Refractory Migraine
Keywords: headache; migraine; lidocaine; glucocorticoid; middle meningeal artery; intra-arterial; status migrainosus
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Lidocaine; Methylprednisolone Hemisuccinate; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): Intra-arterial 80mg lidocaine and 40mg methylprednisolone
  Interventions: Drug: Lidocaine hydrochloride; Drug: Methylprednisolone sodium succinate

INTERVENTIONS:
Drug: Lidocaine hydrochloride — Intra-arterial injection of 40mg lidocaine per middle meningeal artery (total 2 arteries) administered one time
  Other Names: lidocaine; Xylocaine-MPF
Drug: Methylprednisolone sodium succinate — Intra-arterial injection of 20mg methylprednisolone per middle meningeal artery (total 2 arteries) administered one time
  Other Names: methylprednisolone; SOLU-MEDROL

SUMMARY:
The goal of this clinical trial is to test whether injecting lidocaine and steroids into two blood vessels of the brain can help treat chronic headaches (migraines).

The main questions this study aims to answer: is this treatment safe for chronic migraine patients?

Participants will:

* Be treated once with lidocaine and steroid infused into the middle meningeal arteries (two blood vessels in the brain).
* Attend appointments scheduled 1 week, 6 weeks, and 12 weeks after the treatment for a checkup.
* Keep a log of their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 18 years of age.
* Documentation of a diagnosis of intractable migraine without aura, including failure of at least four classes of preventative drugs. Either intolerance or side effects requiring discontinuation or adequate trial at therapeutic dose without relief constitutes failure of therapy.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice contraception during participation in the study. Medically acceptable contraceptives include: (1) surgical sterilization (such as tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants, or injections), (3) barrier methods (such as condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD).
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Patients with concomitant intracranial pathology (e.g., intracranial malignancy).
* Blood glucose level on screening complete metabolic blood panel > 400 mg/dL.
* Patients with known hypersensitivity and/or contraindication to either lidocaine hydrochloride or methylprednisolone sodium succinate, including:
* Patients with known history of hypersensitivity to local anesthetics of the amide type.
* Patients with systemic fungal infections.
* Patients with known or suspected hypersensitivity to cow's milk or its components or other dairy products (SOLU-MEDROL® 40mg presentation includes lactose monohydrate, and may contain trace amounts of milk ingredients).
* Patients taking chronic medications that, when co-administered with lidocaine and other local anesthetics, are at increased risk of developing methemoglobinemia: nitrates/nitrites, local anesthetics, antineoplastic agents, antibiotics, antimalarials, anticonvulsants, acetaminophen, metoclopramide, quinine, sulfasalazine.
* Patients taking chronic medications that, when co-administered with methylprednisolone, are at increased risk for hypokalemia, altered drug levels, convulsions, or altered clearance: amphotericin B, diuretics, aminoglutethimide, macrolide antibiotics, anticholinesterases, antitubercular drugs, cholestyramine, cyclosporine, digitalis glycosides, estrogens (including oral contraceptives), hepatic enzyme inducers/inhibitors, and ketoconazole.
* Patients have known contraindications for angiography. Patients with contrast allergy will be premedicated with diphenhydramine and steroids.
* Patient has known active systemic infection or sepsis.
* Patient has contraindication to anesthetic agents used for conscious sedation/monitored anesthesia care (MAC).
* Concurrent participation in another research protocol for investigation of an experimental therapy.
* Known or suspected inability to adhere to study protocol or protocol requirements, as per the discretion of the Investigator or treating provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | From treatment to 12-week follow-up
  Reported adverse events classified using MedDRA and CTCAE, including all events, treatment-related events, and any serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Tonetti, MD, Principal Investigator — The Cooper Health System; Manisha Koneru, MD, Study Chair — The Cooper Health System; Hamza A Shaikh, MD, Study Chair — The Cooper Health System
Locations (1):
- Cooper University Health Care, Camden, New Jersey, United States

REFERENCES:
- [Result] Koneru M, Shaikh HA, Khalife J, Syrow L, Santucci J, Ballout AA, Patel PD, Thomas AJ, Jovin TG, Tonetti DA. Localized Injection of Lidocaine and Glucocorticoid for Refractory Headache Treatment (LIGHT): A Phase 1 Clinical Trial for Safety. Stroke: Vascular and Interventional Neurology. 2025 Oct 29. https://doi.org/10.1161/SVIN.125.001966

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT06462781/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT06462781/ICF_001.pdf